CLINICAL TRIAL: NCT05057273
Title: A Randomized, Double-Blind Study to Evaluate the Efficacy and Safety of Oral BT-11 in Crohn's Disease Patients With Moderate to Severe Disease
Brief Title: Safety and Efficacy of Oral BT-11 in Crohn's Disease Patients With Moderate to Severe Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision by Landos Biopharma (not related to safety or efficacy)
Sponsor: NImmune Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BT-11-202B
Record Dates: First submitted 2021-08-16; First posted 2021-09-27 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BT-11 880 mg (Experimental): Oral once daily tablet
  Interventions: Drug: BT-11
- Standard of care (Active Comparator): Biologic
  Interventions: Drug: Active comparator

INTERVENTIONS:
Drug: BT-11 — Oral once daily tablet
  Arms: BT-11 880 mg
Drug: Active comparator — Biologic
  Arms: Standard of care

SUMMARY:
This is a phase 2, randomized, double-blind, multicenter study to assess the therapeutic efficacy, safety, and mechanisms of omilancor (BT-11) in patients with moderate to severe Crohn's Disease (CD).

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and female subjects age 18 to 75 years, inclusive.
2. Diagnosis of CD for at least 6 weeks prior to screening
3. Moderate to severely active CD as defined by all of the following:

   * CDAI score of 220-450
   * PRO-2 stool frequency (SF) ≥ 4 and/or abdominal pain (AP) ≥ 2
   * SES-CD ≥ 6 ( ≥4 for isolated ileitis) scored by a blinded central reader

Key Exclusion Criteria:

1. Participant has ulcerative colitis
2. Participant is at imminent risk of ileo-colectomy
3. Prior enrolment in the current study and had received study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Biomarkers of reponse | 12 weeks

IPD SHARING:
Plan to Share IPD: No